CLINICAL TRIAL: NCT04950777
Title: Feasibility and Efficacy of Physical Literacy Screening Integration Into Pediatric Clinical Settings
Acronym: PLAY II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Andrea Stracciolini, Director, Medical Sports Medicine; Attending, Sports Medicine Division, Department of Orthopedic Surgery; Director of Performing Arts Medicine; Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB-P00036957
Record Dates: First submitted 2021-06-29; First posted 2021-07-06 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pediatric ALL; Motility Disorder
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard of care (No Intervention)
- patient education (Experimental): The intervention group will receive the patient education document with their questionnaire, randomization will occur by the study team prior to subject visits. The patient education will be designed to address and investigate the four domains of physical literacy including, knowledge and understanding, motivation and confidence, daily behavior, and physical competence, (i.e., referral based training/PT (passive), self-motivated/directed exercise choice (speaks to child ownership/motivation), simple play outside 60 minutes/day (middle)).
  Interventions: Behavioral: patient education document

INTERVENTIONS:
Behavioral: patient education document — The patient education will be designed to address and investigate the four domains of physical literacy including, knowledge and understanding, motivation and confidence, daily behavior, and physical competence, (i.e., referral based training/PT (passive), self-motivated/directed exercise choice (speaks to child ownership/motivation), simple play outside 60 minutes/day (middle)).
  Arms: patient education

SUMMARY:
The proposed research will be the first study to investigate the feasibility of incorporating physical literacy screening into primary care clinical settings, while determining the efficacy of integration on physical literacy. To investigate aim 1, feasibility, the research team will provide all children ages 6-11 presenting for well-child care by the participating pediatricians with physical literacy screening (PAVSPED) at point of entry for care. The child will complete the 5 yes/no screen and answers will be provided to the pediatrician for acknowledgement. To investigate aim 2, efficacy, participants will be randomized into a control group (standard of care) or an intervention group (patient education). The intervention group will receive the patient education document with their questionnaire, randomization will occur by the study team prior to subject visits. The patient education will be designed to address and investigate the four domains of physical literacy including, knowledge and understanding, motivation and confidence, daily behavior, and physical competence, (i.e., referral based training/PT (passive), self-motivated/directed exercise choice (speaks to child ownership/motivation), simple play outside 60 minutes/day (middle)). All participants will receive a 6-month follow-up email with the same 6 questions to assess if responses changed between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* • Children 6-11 years presenting for an annual well-child appointment at Longwood Pediatrics

Exclusion Criteria:

* • Children with physical handicaps or other significant health problems that would preclude physical activity involvement.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Physical Literacy Vital Sign (PAVSped) total score. | Month 2-4
  Series of yes/no questions surrounding daily moderate to vigorous physical activity. Score is the sum of all positive answers. A higher score means a better outcome, with a minimum value of 0 and maximum value of 5.

SECONDARY OUTCOMES:
Improvement on the follow-up the Physical Literacy Vital Sign (PAVSped) survey total score. | Month 6
  Investigators aim to assess the initial efficacy of PAVSped screening and targeted intervention on the follow-up PAVSped. The score is the sum of all positive answers. A higher score means a better outcome, with a minimum value of 0 and maximum value of 5.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Stracciolini, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
All data will be handled by IRB approved staff. The numerical code used to identify subjects will be kept separately in a password-protected file and will not be accessible from the rest of the database. All patient information will be stored within the Boston Children's server within a locked departmental folder. Patient data will be entered into REDCap by the patients filling out the questionnaire. No information will be kept on personal computers.